CLINICAL TRIAL: NCT04877418
Title: Tele-rehabilitation Through Constraint Induced Movement Therapy (TeleCIMT) at Recovering the Function of the Upper Limb and Quality of Life
Brief Title: Tele-rehabilitation Through CIMT at Recovering the Function of the Upper Limb and Quality of Life
Acronym: TeleCIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, ARLETTE PATRICIA DOUSSOULIN SANHUEZA, Principal Investigator, Universidad de La Frontera
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIUFRO
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Telerehabilitation
Keywords: Telerehabilitation; Constraint Induced Movement therapy; Upper limb; Outcomes; Functionality; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TeleCIMT group (Experimental): One month after baseline evaluations, patients will receive a 3-week program through TeleCIMT.
  * Task Oriented Repetitive Training
  * Use of the Affected Upper Extremity
  * Transfer Package
  Interventions: Procedure: TeleCIMT

INTERVENTIONS:
Procedure: TeleCIMT — Mode applied remotely, through the principles and components of the CIMT protocol.

SUMMARY:
The current pandemic scenario is immensely challenging for healthcare professionals. Telerehabilitation,is a promising option that benefited many people, allowing continuity of therapeutic processes and promoting the admission of people without prior access to rehabilitation programs. This modality has shown comparable results with conventional rehabilitation strategies, applied in patients with neurological pathologies. However, the modalities applied and the quality of the studies are insufficient to establish their real benefits and effectiveness.

Strategies such as CIMT, have been shown to be effective in improving upper limb function and restoring quality of life in stroke survivors. However, there is little evidence on its effectiveness when administered under telerehabilitation modality.

DETAILED DESCRIPTION:
Objective To determine if movement-induced restriction therapy, delivered through telerehabilitation (TeleCIMT), recovers function and improves quality of life in patients with brachial sequelae, after a stroke.

Methodology A prospective, single-group experimental study will be conducted. The sample will be of an intentional type, selected according to meeting the inclusion criteria. Each participant will be evaluated three times, at the beginning, middle and end of the intervention using TeleCIMT. The evaluation scales to be used will be Motor Activity Log-30 (MAL-30) and Action Research Arm for function and ECVI-38 scale for quality of life. The difference between these measurements in each patient (change score) will express the progress (or setback) obtained through this modality of intervention via telerehabilitation. Specifically, the effects of the TeleCIMT will be examined by one-factor within-subject analysis of variance (ANOVA) using time (T1, T2, and T3) as the independent variable and the recovery measures as dependent variables. In all analyzes, results with p values less than or equal to 0.05 will be considered statistically significant.

Expected results Through this proposal, the aim is to promote a line of research that allows the development of scientific evidence in the area of telerehabilitation in subjects with neurological pathologies. This information will benefit numerous professionals, promoting timely access to rehabilitation, providing continuity in therapeutic processes and reversing levels of disability due to neurological pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 30 and 80 years.
* Who present a single stroke event confirmed by CT,
* Between 5 and 14 points on the NIHSS Scale
* Who have the ability to sit independently.
* Who can follow simple instructions (score greater than 13 on the Mini Menta)l.
* <2 points on the Modified Ashworth Scale on elbow and wrist
* <4 points on the Visual Analog Scale on shoulder.
* That they can perform a functional test of 20 ° of wrist extension and 10 ° of finger extension (take and drop a cloth with the affected hand).

Exclusion Criteria:

* Severe cognitive impairment (aphasia, attention deficit, reasoning or memory disorders).
* Severe sensory impairment (visual-auditory).
* Orthopedic limitation (use of a cane).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Upper limb function in patients after stroke. | 3 weeks
  MAL: It is a structured interview, composed by 30 items, intended to examine how much and how well the subject uses their more-affected arm outside of the laboratory setting. During the test administration. participants should be told that they can give half scores (i.e., 0.5,1.5,2.5,3.5,4.5) if this is reflective of their ratings.
  ARAT: It is a performance test that evaluates the ability of the affected upper limb to pick up, move and grasp objects of different size, weight and shape in patients with cortical injury. It is composed of 19 items that examine grip, grip, clamp and gross movement. The total score ranges from 0 (none of the movements were performed) to 57 (all the movements were performed without difficulty).
  The application of both instruments will be carried out virtually according to standardized procedures.

SECONDARY OUTCOMES:
The quality of life of patients after stroke. | 3 weeks.
  It will be evaluated through the ECVI-38 scale, which comprises 38 items grouped into 8 subscales: physical state, communication, cognition, emotions, feelings, basic activities of daily life, common activities of daily life and socio-family functioning. It also contains two additional questions about sexual relationships and work activity. The application will be carried out virtually according to standardized procedures in the manual.
  The formulation of responses is with a Likert scale, from 5 to 1, where 5 is the worst score as evaluated and 1 is where the patient reports having no difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Arlette Doussoulin, PHD, Principal Investigator — Universidad de La Frontera
Locations (1):
- Universidad de La Frontera, Temuco, Chile

IPD SHARING:
Plan to Share IPD: No
The research team is in talks with their counterpart from the University of Sydney, led by Dr. Lauren Christie, who are developing research on the same topic of study.